CLINICAL TRIAL: NCT06611371
Title: A Phase I/II, Observer-Blind, Randomized, Placebo-Controlled, Dose-Selection Study to Assess the Safety, Tolerability, and Immunogenicity of Hexavalent Group B Streptococcus Conjugate Vaccine Manufactured by Inventprise, Inc., in Healthy, Non-Pregnant, Adult Women of Childbearing Age (WOCBA) in the US and South Africa.
Brief Title: Phase I/II Study to a Assess the GBS-06 Vaccine Manufactured by Inventprise, Inc., in Healthy, Non-Pregnant, Adult Women of Childbearing Age.
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inventprise Inc. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 103
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Group B Streptococcal Infections
Keywords: Group B streptococcus (GBS); Vaccine; Healthy Volunteer
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Intervention Model Description: Single dose of low, mid or high concentrations of IVT GBS-06, or a placebo (saline control) at Day 1 (Randomized 1:1:1:1). The four study groups will be enrolled simultaneously to allow for parallel assessments of participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects randomized 1:1:1:1, placebo-controlled, observer blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1; GBS-06 (Low) (Experimental): Participants will receive a single 0.5mL dose of IVT GBS-06 Formulation 1 (low dose polysaccharide concentration) administered by intramuscular injection to the non-dominant deltoid muscle on Day 1.
  Interventions: Biological: IVT GBS-06
- Group 2; GBS-06 (Mid) (Experimental): Participants will receive a single 0.5mL dose of IVT GBS-06 Formulation 2 (mid-dose polysaccharide concentration) administered by intramuscular injection to the non-dominant deltoid muscle on Day 1.
  Interventions: Biological: IVT GBS-06
- Group 3; GBS-06 (High) (Experimental): Participants will receive a single 0.5mL dose of IVT GBS-06 Formulation 3 (high dose polysaccharide concentration) administered by intramuscular injection to the non-dominant deltoid muscle on Day 1.
  Interventions: Biological: IVT GBS-06
- Group 4; Placebo (Placebo Comparator): Participants will receive a single 0.5mL dose of 0.9% sodium chloride placebo administered by intramuscular injection to the non-dominant deltoid muscle on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IVT GBS-06 — Hexavalent Group B Streptococcus polysaccharide conjugate vaccine (serotypes Ia, Ib, II, III, V, and VII) administered as a single dose.
  Arms: Group 1; GBS-06 (Low); Group 2; GBS-06 (Mid); Group 3; GBS-06 (High)
Biological: Placebo — 0.9% sodium chloride
  Arms: Group 4; Placebo

SUMMARY:
To assess the safety and tolerability of IVT GBS-06 vaccine administered as a single-dose regimen, at three dosage levels in healthy, non-pregnant, adult women of childbearing age (WOCBA).

DETAILED DESCRIPTION:
This is a phase I/II, randomized, placebo-controlled, observer-blinded trial to evaluate the safety, tolerability, and immunogenicity of a multivalent GBS vaccine candidate in healthy, non-pregnant, adult WOCBA, 18-49 years of age, at two sites, one each in the US and South Africa. Approximately 600 participants will be randomized to receive a single dose of low, mid, or high concentration of IVT GBS-06, or a placebo (saline control) at Day (D)1, administered IM by injecting 0.5 mL into the deltoid muscle. The three dose levels denote the amount of capsular polysaccharide (CPS) for each of the six serotypes per 0.5 mL. These four study groups will be enrolled simultaneously to allow for parallel assessments of overall IVT GBS-06 safety and tolerability. Participants will be randomized in a 1:1:1:1 ratio to one of the dose levels or placebo. This study will utilize a sentinel-cohort design in which 20 participants overall (i.e., N=5 per treatment arm) at the US site will be randomized, vaccinated, and evaluated for safety prior to opening enrolment of additional participants in USA and in South Africa. This study targets representation from both study populations and therefore at least 220 participants will be recruited from each of the two sites and will allow competitive enrollment across the two study sites for the remaining 160 participants to reach 600 within target enrollment period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women aged 18-49 years (inclusive) at enrollment.
2. Healthy, as defined by the absence of any clinically significant medical conditions, either acute or chronic, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator. Participants with stable chronic conditions may be enrolled in the study at the discretion of the investigator. Stable conditions are conditions that do not require changes to medication or other interventions in the past 6 weeks.
3. Willing and able to provide written informed consent prior to performance of any study specific procedure.
4. If of childbearing potential*, not be breastfeeding and not be pregnant (based on a negative serum pregnancy test at screening and a negative urine pregnancy test during the 24 hours prior to study vaccination) and having practiced adequate contraception** for at least 30 days prior to study vaccination and willing to continue using adequate contraception consistently throughout the study.

   * Participants can be considered not of childbearing potential if they meet at least 1 of the following criteria:

     * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state.
     * Have undergone a documented hysterectomy and/or bilateral oophorectomy.
     * Have medically confirmed ovarian failure.
     * They identify as transgender women and do not have ovaries or a uterus. All other participants (including participants with tubal ligations) are considered to be of childbearing potential.

       ** Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example:
     * Abstinence from penile-vaginal intercourse
     * Combined estrogen and progesterone oral contraceptives
     * Hormonal (e.g., progestogen) injections
     * Hormonal (e.g., etonogestrel or levonorgestrel) implants
     * Contraceptive vaginal ring
     * Percutaneous contraceptive patches
     * Intrauterine device
     * Intrauterine hormonal system
5. Resides in the study area and is able and willing to adhere to all study restrictions and to all study visits and procedures including completion of seven day post-injection memory aid (as evidenced by a signed informed consent form and assessment by the investigator).

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from participation:

1. Presence of an acute disease within 72 hours prior to enrollment - temporary exclusion*.
2. Presence of recorded fever (axillary temperature ≥ 37.5°C or oral temperature of ≥ 37.5°C) or use of an antipyretic medication within 72 hours prior to enrollment- temporary exclusion *.
3. Presence of an abnormal (> Grade 2) vital sign measurement (heart rate, blood pressure[systolic or diastolic], respiratory rate) - temporary exclusion*
4. Laboratory confirmed active infection with human immunodeficiency virus, chronic hepatitis B virus infection (hepatitis B virus surface antigen positive), or hepatitis C virus infection. HCV RNA negative (if tested) may be allowed.
5. BMI <17 or ≥ 40 kg/m2
6. Presence of any chronic or degenerative neurological disease or history of significant neurological disorder (e.g., dementia, meningitis, seizures, multiple sclerosis, vasculitis, or Guillain-Barré syndrome), genetic/congenital or acquired.
7. Evidence of a major depression disorder not well controlled in the past 2 years prior to screening (by history and medication review, at discretion of the investigator) or history of suicidal ideation or attempt in the past 2 years prior to screening.
8. History of severe adverse reaction and/or severe allergic reaction (e.g., anaphylaxis) to polyethylene glycol (PEG) or any vaccine.
9. History of microbiologically proven invasive disease caused by GBS (S. agalactiae) or receipt of any investigational GBS vaccine.
10. Participation in another investigational product (drug or vaccine) clinical trial within 30 days prior to enrollment in this study or receipt of any such investigational product other than the study vaccine within 30 days prior to administration of study vaccine or planned use during the study period.
11. Immunocompromising condition with known or suspected immunodeficiency.
12. Prior use of or anticipated need of any long-acting immunomodulating drug (e.g., infliximab or rituximab cytotoxic agents), or chronic administration (defined as more than 14 days) of high dose (≥ 20 mg of prednisolone or equivalent/day) systemic corticosteroids during the study period. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 30 days before investigational product administration. Inhaled/nebulized, intra-articular, intra-bursal, or topical (skin or eyes) corticosteroids are permitted.
13. Indications of drug abuse or excessive use of alcohol as deemed by the investigator to confound safety assessments or render the participant unable or unlikely to adhere to protocol requirements or provide accurate safety reports.
14. Administration of any vaccine other than the study vaccine within 28 days prior to or after study vaccination. Exceptions of seasonal inactivated influenza and COVID-19 vaccines which are prohibited for only 14 days prior to or following study vaccination is applicable.
15. Receipt of transfusion of any blood product or application of immunoglobulins within the 12 weeks prior to the administration of study vaccine or planned use during the study period.
16. Any planned surgery during the study period that would require hospitalization, use of prohibited medication, or will interfere with follow-up visits.
17. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding.
18. Participant is an employee of, or close personal relation of any person employed by the Sponsor, PATH, the CRO, the PI, or key study site personnel.
19. History of malignancy, excluding non-melanoma skin and cervical carcinoma in situ.
20. Any other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for enrollment into this study.
21. Any screening laboratory value that meets the criteria specified below will be excluded from study participation:

    1. Hemoglobin < 10.0 g/dL.
    2. White blood cells (WBC) increased > 15,000 cells/mm3
    3. WBC decreased < 2,600 cells/L
    4. Platelet count < 125,000 cells/mm3
    5. Creatinine >1.8 mg/dL or 159.1 µmol/L
    6. Alanine aminotransaminase (ALT) > 2.5 × the upper limit of normal (ULN)
    7. Total bilirubin > 1.5 × ULN

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women between the ages of 18 to 49.
Enrollment: 600 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety -percentage of participants reporting immediate AE within 30 minutes of vaccination | 30 minutes after vaccination
  The percentage of participants reporting immediate AE within 30 minutes of vaccination.
Safety - percentage of participants reporting solicited local adverse events (AEs) within 7 days of vaccination | Day 1 - Day 7 after vaccination
  The percentage of participants reporting solicited local adverse events (AEs) within 7 days following study vaccination (pain, redness and swelling/induration at the injection site).
Safety- percentage of participants reporting solicited systemic AEs within 7 days following study vaccination (fever, fatigue, headache, chills, myalgia, arthralgia, and nausea/vomiting) | Day 1 - Day 7 after vaccination
  The percentage of participants reporting solicited systemic AEs within 7 days following study vaccination (fever, fatigue, headache, chills, myalgia, arthralgia, and nausea/vomiting)
Safety - percentage of participants reporting unsolicited AEs within 28 days following study vaccination | Day 1 - Day 28 after vaccination
  The percentage of participants reporting unsolicited AEs within 28 days following study vaccination
Safety - percentage of participants with clinically significant laboratory abnormalities within 7 days following study vaccination | Day 1 - Day 7 after vaccination
  The percentage of participants with clinically significant laboratory abnormalities within 7 days following study vaccination
Safety - percentage of participants reporting medically attended adverse events (MAAEs) | From Day 1 vaccination through the end of study
  The percentage of participants reporting medically attended adverse events (MAAEs)
Safety - percentage of participants reporting serious adverse events (SAEs) | From Day 1 vaccination through the end of study
  The percentage of participants reporting serious adverse events (SAEs)

SECONDARY OUTCOMES:
Immunogenicity - IgG | Day 1 baseline collection through 4-weeks post dose collection
  Percentage of participants that seroconvert per serotype. Seroconversion is defined as induction of a serotype-specific anti- capsular polysaccharide (anti-CPS) IgG concentration that is at least 4-fold greater than the Multiplex immunoassay (MIA) lower limit of quantitation (LLOQ) or the baseline level, whichever is higher.
Immunogenicity - IgG | Day 1 baseline collection and 4-weeks post dose collection
  Percentage of participants attaining or exceeding a concentration of 0.2, 0.5, 1 and 2 µg/mL of serotype-specific IgG. The rate will be assessed overall and stratified by baseline seropositivity.
Immunogenicity - IgG | Day 1 baseline collection and 4-weeks post dose collection
  Geometric mean concentration (GMC) of GBS-06 serotype specific IgG
Immunogenicity - IgG | Day 1 baseline collection and 4-weeks post dose collection
  Geometric mean fold-rise (GMFR) of GBS-06 serotype specific IgG
Immunogenicity - IgG | Day 1 baseline collection and 4-weeks post dose collection
  Rank of IVT GBS-06 dosage levels according to the serotype-specific seroconversion percentages and GMFR
Immunogenicity - IgG | Day 1 baseline collection and 4-weeks post dose collection
  Difference in serotype-specific seroconversion percentage for each IVT GBS-06 dosage level and placebo.
Immunogenicity - IgG | Day 1 baseline collection and 4-weeks post dose collection
  Difference in percentage of participants attaining or exceeding a concentration of 0.2, 0.5, 1, and 2 µg/mL of serotype specific IgG for each IVT GBS-06 dosage level and placebo.
Immunogenicity | Day 1 baseline collection and 4-weeks post dose collection
  GMC serotype-specific ratio between each IVT GBS-06 dosage level and placebo.
Immunogenicity | Day 1 baseline collection and 4-weeks post dose collection
  GMFR serotype-specific ratio between each IVT GBS-06 dosage level and placebo.
Immunogenicity - OPA | Day 1 baseline collection and 4-weeks post dose collection
  Post vaccination IVT GBS-06 serotype specific OPA geometric mean titer (GMT) assessed overall and stratified by baseline seropositivity. OPA seropositivity cut off will be based on LLOQ for each serotype calculated in µg/ml.
Immunogenicity - OPA | Day 1 baseline collection and 4-weeks post dose collection
  IVT GBS-06 serotype-specific OPA GMFR from baseline
Immunogenicity - OPA | Day 1 baseline collection and 4-weeks post dose collection
  IVT GBS-06 serotype-specific OPA GMT ratio between each IVT GBS-06 level and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Tasker, MD, MPH, FIDSA, Study Director — Inventprise Inc.
Locations (2):
- NYU Grossman School of Medicine, New York, New York, United States
- Wits Vaccines and Infectious Diseases Analytics Research Unit (Wits-VIDA), University of the Witwatersrand, Johannesburg, Gauteng, South Africa